CLINICAL TRIAL: NCT02656862
Title: Causes of Acute Undifferentiated Fever in Outpatients in the Democratic Republic of Congo
Acronym: RESFANDI
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Universiteit Antwerpen (Other); University of Kinshasa (Other)
Responsible Party: Sponsor
Other Study IDs: RESFANDI
Record Dates: First submitted 2016-01-05; First posted 2016-01-15 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Undifferentiated Acute Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
Fever is one of the main reasons for outpatient consultations in sub-saharan Africa. Following the introduction of malaria RDTs, clinicians face a high number of malaria-negative patients for whom they do not have a clear diagnosis. Through clinical history and examination, acute fever patients are categorized into: acute respiratory infections, urinary tract infections and other focal infections, diarrheal fevers and undifferentiated fevers. The latter being patients where no focal source of infections can be found during the consultation visit. In this proposal, the investigators focus on these acute undifferentiated fevers in an outpatient clinic.

These fevers have the challenge of few point-of-care tests (POCT) available for the clinicians to identify the etiology of fever and guide treatment in resource-limited countries. As a consequence, over-prescription of antibiotics has increased. In order to improve patient outcomes while supporting judicious use of antimicrobials, there is an urgent need to change the management of febrile patients in low-income countries. This can only be achieved by providing evidence-based clinical guidelines for the management of these acute febrile patients. To develop such guidelines, epidemiological data on etiologies of undifferentiated fever need to be generated. The investigators will evaluate pathogen infection (such as dengue, chikungunya and others) in 640 patients ≥ 2 years old with acute undifferentiated fever. To evaluate the existence of aspecific and subclinical infections and co-infections, the investigators will also test a subsample of 200 patients with ARI, UTI, diarrheal fever and malaria. The investigators expect to have as main results: proportions of each syndrome among fever patients, key pathogens associated with undifferentiated fever and their clinical presentation and demographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 years old
* a history of acute fever (i.e. ≥ 2 days and ≤ 7 days)
* an axillary temperature of ≥37.5°C
* written informed consent obtained;

Exclusion Criteria:

* main complaint for consultation is an injury, trauma or poisoning
* hospitalization or delivery in the preceding 2 weeks
* suspicion of meningitis/encephalitis

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will take place in the Lisungi Health centre, Pumbu. Pumbu is a health area of about 14 000 inhabitants, belonging to the municipality of peri-urban Mont Ngafula 1, at the southern side of Kinshasa. The Lisungi health centre is the only public health facility in the health area, with on average 250 consultations/week. About 70% of attending patients have fever as reason for consultation.
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of key pathogens among study participants with 'undifferentiated fever' | At consultation over a period of 6 months
  The key pathogens will be identified through specific laboratory diagnostic tests on the blood/serum of included patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Lutumba, PhD, Principal Investigator — Institut National de Recherche Biomédicale (INRB), Kinshasa
Locations (1):
- Lisungi Health Center, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Proesmans S, Katshongo F, Milambu J, Fungula B, Muhindo Mavoko H, Ahuka-Mundeke S, Inocencio da Luz R, Van Esbroeck M, Arien KK, Cnops L, De Smet B, Lutumba P, Van Geertruyden JP, Vanlerberghe V. Dengue and chikungunya among outpatients with acute undifferentiated fever in Kinshasa, Democratic Republic of Congo: A cross-sectional study. PLoS Negl Trop Dis. 2019 Sep 5;13(9):e0007047. doi: 10.1371/journal.pntd.0007047. eCollection 2019 Sep. PMID 31487279